CLINICAL TRIAL: NCT06816901
Title: Measuring Lactation Initiation After Early Postpartum Injectable Progestin (DMPA) Use Among Women in Dhanusha District of Nepal: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Center for Research on Environment, Health and Population Activities (Other)
Responsible Party: Principal Investigator, Sarah Averbach, MD MAS, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 811161
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Contraception; Depot Medroxyprogesterone Acetate; Lactation; DMPA
Keywords: Depo; Injectable contaception; postpartum; contraception; family planning; DMPA
MeSH Terms: conditions — Breast Feeding | interventions — Medroxyprogesterone Acetate; N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Initiation of injectable depo medroxyprogesterone acetate (DMPA) within 48 hours of birth
  Interventions: Drug: Depo Medroxyprogesterone acetate

INTERVENTIONS:
Drug: Depo Medroxyprogesterone acetate — Initiation of injectable depo medroxyprogesterone acetate (DMPA) contraception within 48 hours after birth
  Other Names: DMPA; Injectable contraception

SUMMARY:
This is a pilot study of early postpartum initiation of the injectable progestin contraception, depo medroxyprogesterone acetate (DMPA), among 40 postpartum people. The study aims to assess the feasibility to conduct a larger trial evaluating the effects of early postpartum initiation DMPA on lactation and infant growth outcomes in Nepal.

DETAILED DESCRIPTION:
The primary objective of this study is to pilot the procedures necessary to demonstrate feasibility for a larger randomized trial evaluating the effects of early postpartum initiation of DMPA on time to lactogenesis (transition to mature milk), lactation continuation, and infant growth and development.

The investigators will conduct a pilot study among 40 birthing people who deliver a singleton, healthy, term infant; intend to feed their infant human milk (breastfeed) exclusively for at least 6 months; and plan to use DMPA for postpartum contraception. Participants will be administered DMPA within 48 hours after birth and will be followed for 12 weeks postpartum. Time to lactogenesis, the proportion of participants exclusive feed their infant human milk at 12 weeks, any lactation and infant growth through 12 weeks will be measured. We will analyze time to onset of lactogenesis the proportion of participants exclusively feeding human milk at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Currently live in Nepal
* Had a vaginal or cesarean delivery of a singleton full-term infant within the past 48 hours
* Not yet undergone lactogenesis
* Desire to use DMPA as a method of postpartum contraception

Exclusion Criteria:

* Desire a repeat pregnancy in less than 6 months
* Do not intend to exclusively feed infant own human milk for 6 months
* Do not have access to a telephone
* Any medical contraindication to DMPA
* Any contraindication to human milk feeding for their infant
* History of breast surgery (augmentation or reduction)
* Infant with a major congenital anomaly (will be excluded due to unique challenges with feeding in these populations)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Enrollment feasibility | 12 weeks
  The ability of project staff to consent and enroll 40 individuals who are willing to participate in this pilot study within 12 weeks.

SECONDARY OUTCOMES:
Time to lactogensis | 148 hours
  Amount of time (in hours) from birth to lactogenesis
Exclusive lactation | 12 weeks
  Proportion of participants who report exclusive lactation without supplementation
DMPA Continuation | 12 weeks
  The proportion of participants who use DMPA continuously for 12 weeks and return for a second dose
Change in infant weight | Birth to 4 weeks
  Infant weight in grams will be compared over 4 weeks
Change in infant length | Birth to 4 weeks
  Infant length in millimeters will be compared over 4 weeks
Change in infant head circumference | Birth to 4 weeks
  The maximum diameter through the infant's glabella and occiput is found and measured with a tape measure and recorded to the nearest millimeter and compared over 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Averbach, MD, MAS, Principal Investigator — University of California, San Diego
Locations (1):
- Provincial Hospital Janakpur of Dhanusha district, Janakpur Dham, Dhanusha District, Nepal

IPD SHARING:
Plan to Share IPD: No